CLINICAL TRIAL: NCT00032539
Title: CSP #476CC - Enhancing Quality of Informed Consent (EQUIC-CC) Customized Consent
Brief Title: EQUIC-CC: Enhancing Quality of Informed Consent - Customized Consent
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 476CC
Record Dates: First submitted 2002-03-27; First posted 2002-03-28 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: Informed Consent

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
Patients in 'parent' cooperative study projects are interviewed about their experiences in the informed consent process.

DETAILED DESCRIPTION:
Intervention: (1) Cognitive stratification (obtained by a test of cognitive ability, followed by a tailored IC process); (2) Pre-recruitment video (a patient-activation video designed to prevent several common misconceptions; (3) Provide prospective research volunteers with a sense of the purpose and methods of controlled research); and (4) Evaluation of the informed consent process using the Brief Informed Consent Evaluation Protocol (BICEP) developed in EQUIC-DP.

Primary Hypothesis: The validity of informed consent can be improved, as measured by an independent interview of patients (BICEP), by at least one of three interventions described above.

Primary Outcomes: The quality of the informed consent process, as measured by the BICEP (Brief Informed Consent Evaluation Protocol). The BICEP also offers a method to certify informed consent in routine use.

Study Abstract: Customized Consent will develop and test an innovative, supplemental method of disclosing information to patients in the informed consent process. This disclosure strategy is intended to increase patients' understanding and satisfaction with the consent process. This study has two goals:

* to evaluate the effectiveness of an intervention to improve comprehension during informed consent; and
* to identify those patients for whom this intervention is most effective.

The primary goal of EQUIC-CC is to determine whether an intervention, added to usual procedures for obtaining informed consent, is able to improve comprehension. The second goal of EQUIC-CC is to identify those patients for whom an augmented consent intervention is most effective, as well as to determine which subgroups of patients, if any, are most likely to benefit from visual information added to the usual disclosure phase of obtaining informed consent.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Depends on 'parent' study

Exclusion Criteria:

Exclusion Criteria:

* Depends on 'parent' study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Veterans in selected clinical trials conducted by VA
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 1999-04; Primary Completion 1999-04 (Actual); Study Completion 1999-04 (Actual)

PRIMARY OUTCOMES:
improve method of disclosing information to patients in the informed consent process | post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Philip Lavori, PhD, Study Chair — Stanford University
Locations (4):
- United States (4):
  - VA Palo Alto Health Care System, Palo Alto, California
  - Stanford University, Stanford, California
  - VA Medical Center, Durham, Durham, North Carolina
  - VA Medical Center, Philadelphia, Philadelphia, Pennsylvania